CLINICAL TRIAL: NCT06148987
Title: Reliability and Validity of the Turkish Version of the Smart Tools Proneness Questionnaire
Brief Title: Turkish Version of the Smart Tools Proneness Questionnaire
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Assoc. Prof., Çankırı Karatekin University
Other Study IDs: ab2e5654208645eb
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Health, Subjective
Keywords: Smart Devices; Human-Tool Interaction; Reliability and Validity; Digital Literacy
MeSH Terms: interventions — Surveys and Questionnaires; Demography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire group: This study will be conducted in Turkey between January and August Ferbruary 2024, and it aims to investigate the Turkish translation, reliability, and validity of the AAE-A survey. All participants must meet the following inclusion criteria: (i) be 18 years old or older, (ii) use smart devices and tools, and (iii) provide written consent to participate. Participants with specific abnormalities such as cognitive or neurological disorders, upper extremity pain, functional limitations, or cognitive impairments will be excluded from the study to ensure the accuracy of the norms. It is estimated that a sample size of 270 individuals, with 10 individuals per item, will be needed for the sample size of this study."
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The translation and cultural adaptation of the survey will be conducted according to the guidelines of Beaton et al. Following the Beaton guidelines, the translation and cultural adaptation steps are as follows: 1) The original version of the survey will be translated into Turkish separately by two individuals whose native language is Turkish and who are proficient in English. One translator will be an English linguistics scholar unfamiliar with the concepts and terms, while the other will be a physiotherapist familiar with the concepts and terms; 2) Subsequently, the translations will be merged into a single text by these two translators; 3) The final Turkish version of the survey will be translated back into English by two translators who are unaware of the study; 4) The translations will then be combined by these two translators to create a harmonized and single text; 5) The back-translation and cultural adaptation
  Other Names: Demographic Data

SUMMARY:
Technologically advanced tool solutions (i.e., the highest level of automation) may not always be the preferred choice for participants when given an option. Various experiments show that in vehicles, low to moderate levels of automation are often preferred over highly automated vehicles. The association of higher task demands with smarter tools has been reported to influence tool selection along with task demand. However, participants may avoid using a fully automatic tool even if the task is highly laborious. In fact, in a series of experiments, participants more distinctly preferred manually completing routine tasks over more efficient fully automatic task completion.

Based on these collective theories, the Smart Tools Proneness Questionnaire (STP-Q), developed by Navarro J. and colleagues, aims to explore and measure interindividual differences influencing an individual's propensity to use smart tools, their initial selection of smart tools, and subsequent usage. In practice, measuring the propensity of any individual to use smart tools will be significantly beneficial for both professionals and non-professionals involved in designing, producing, and implementing such tools. Therefore, the purpose of this study is to translate, validate, and establish the reliability of the Turkish version of the STP-Q.

DETAILED DESCRIPTION:
Individuals have developed a unique and enduring relationship with the tools they use. This relationship can be described as the creation and use of tools to define the human species. With advancements in techniques and technologies, complex human-tool interactions now occur in many daily situations. The development of these more complex human-tool interactions accompanies the creation of smarter tools. These advanced tools are increasingly inclined towards autonomy and their functionalities now surpass the understanding of most users, and even the initial designers.

Smart tools are understood as any machine or device that can complete tasks involving information, mechanics, or electronics in lieu of or in connection with individuals. The smartphone can now be considered a ubiquitous example of such tools, reaching approximately half or more of the global population in the past decade. In high-income countries in North America and Europe, over 80% of the population owns a smartphone. The idea that individual differences play a crucial role in the implementation of any technological innovation has become a recurring theme in various disciplines, including information systems, manufacturing, and marketing.

Technologically advanced tool solutions (i.e., the highest level of automation) may not always be the preferred choice for participants when given an option. Various experiments show that in vehicles, low to moderate levels of automation are often preferred over highly automated vehicles. The association of higher task demands with smarter tools has been reported to influence tool selection along with task demand. However, participants may avoid using a fully automatic tool even if the task is highly laborious. In fact, in a series of experiments, participants more distinctly preferred manually completing routine tasks over more efficient fully automatic task completion.

Based on these collective theories, the Smart Tools Proneness Questionnaire (STP-Q), developed by Navarro J. and colleagues, aims to explore and measure interindividual differences influencing an individual's propensity to use smart tools, their initial selection of smart tools, and subsequent usage. In practice, measuring the propensity of any individual to use smart tools will be significantly beneficial for both professionals and non-professionals involved in designing, producing, and implementing such tools. Therefore, the purpose of this study is to translate, validate, and establish the reliability of the Turkish version of the STP-Q.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for participants in this validation study require individuals to be 18-55 years, actively use smart devices, provide written consent, possess proficiency in the Turkish language, and not have specific abnormalities or impairments that may hinder accurate survey completion. Ethical considerations, aligned with the principles of the Helsinki Declaration, will be maintained throughout the study.

Exclusion Criteria:

* Conversely, exclusion criteria involve disqualifying individuals below the age of 18 or above 55, non-users of smart devices, those unwilling to provide written consent, individuals lacking proficiency in Turkish, and those with physical or cognitive impairments. This comprehensive approach ensures that participants are suitable for the research, promoting reliable and meaningful responses while upholding ethical standards in the study's execution.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  * The inclusion criteria for participants in this validation study require individuals to be 18-55 years, actively use smart devices, provide written consent, possess proficiency in the Turkish language, and not have specific abnormalities or impairments that may hinder accurate survey completion. Ethical considerations, aligned with the principles of the Helsinki Declaration, will be maintained throughout the study.
  Exclusion Criteria:
  * Conversely, exclusion criteria involve disqualifying individuals below the age of 18 or above 55, non-users of smart devices, those unwilling to provide written consent, individuals lacking proficiency in Turkish, and those with physical or cognitive impairments. This comprehensive approach ensures that participants are suitable for the research, promoting reliable and meaningful responses while upholding ethical standards in the study's execution.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Smart Tool Proneness Qustionnaire | 15 Minutes
  The Smart Tool Proneness Qustionnaire (STP-Q): STP-Q is a 27-item self-report scale that assesses an individual's inclination to use smart devices on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). The total score of the scale ranges from 27 to 189, where a higher score indicates a stronger inclination. STP-Q provides practitioners with an individual tendency measure in three dimensions of using smart devices: utilitarian use, hedonic and social use, and inclination to delegate tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)